CLINICAL TRIAL: NCT01898559
Title: Nicotine Metabolism and Little Cigars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 816605
Record Dates: First submitted 2013-07-03; First posted 2013-07-12 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Smoking
Keywords: little cigars; cigarettes; smoking
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Black & Mild little cigars (Experimental): Participants switch from smoking their own brand of cigarettes to only smoking Black & Mild little cigars.
  Other: Switch to smoking only little cigars
  Interventions: Other: Switch to smoking only little cigars
- King Edward little cigars (Experimental): Participants switch from smoking their own brand of cigarettes to only smoking King Edward little cigars.
  Other: Switch to smoking only little cigars
  Interventions: Other: Switch to smoking only little cigars

INTERVENTIONS:
Other: Switch to smoking only little cigars — Participants smoke only little cigars for 15 days.

SUMMARY:
This study examines the effects of smoking little cigars in different groups of smokers. The investigators are focusing on differences in how smokers' bodies break down and eliminate nicotine from their systems. Some people are fast metabolizers of nicotine, meaning they break down and eliminate nicotine from their bodies more quickly. Other people are slower metabolizers meaning they break down and eliminate nicotine more slowly. The investigators are comparing these two groups of smokers when they switch to smoking cigars instead of cigarettes.

DETAILED DESCRIPTION:
This study examines the effects of switching from cigarette to little cigar smoking on smoking behaviors and toxin exposure in fast and slow nicotine metabolizing smokers. We will recruit current smokers (split between slow and rapid nicotine metabolizing smokers) for a 20-day protocol. Participants will smoke their own brand cigarettes during a baseline 5 day period, followed by 15 days smoking little cigars. This study will use a validated, phenotypic marker of nicotine metabolism rate that may identify those individuals at greatest risk of harm exposure when using little cigars. This study will examine the compensatory effects of little cigars on smoking behaviors and toxin exposure among slow and rapid nicotine metabolizers.

ELIGIBILITY:
Inclusion Criteria:

* adults age 21-65.
* smoking at least 10 cigarettes per day.
* smoking daily for the last 5 years.
* Provide a baseline breath CO reading 10 parts per million.
* smoke predominantly filtered cigarettes.
* not currently using any other nicotine containing products such as smokeless tobacco, nicotine
* replacement therapies (patch or gum).
* are fluent in English and are capable of providing written informed consent, which includes compliance with the requirements and restrictions listed in the combined consent and HIPAA form.
* Have smoked at least 25 cigars in their lifetime
* Participants who meet the inclusion/exclusion criteria and attend an Intake Visit for medical screening will be asked to provide a blood sample to determine NMR. Only those individuals who are characterized as slow or rapid, based on NMRs .26, or .42, will be eligible.

Exclusion Criteria:

1. use of any nicotine containing products other than cigarettes
2. current or impending enrollment in smoking cessation program
3. history in the last year or current treatment of substance abuse (other than nicotine dependence)
4. positive drug screen for cocaine or opiates for urine drug screen at intake session
5. alcohol use greater than 25 standard drinks per week
6. current or planned pregnancy or lactating
7. history or current diagnosis of psychosis, bipolar disorder, mania, or schizophrenia
8. current major depression (history of major depression but in remission for a minimum 6 months is eligible).
9. serious or unstable disease within past year (e.g. cancer other than melanoma, heart disease)
10. history or current diagnosis of COPD
11. history of stroke or heart attack
12. age less than 21 years- participants must be 21 years old to give consent to volunteer
13. age more than 65 years - smoking is often associated with cardiovascular and pulmonary obstructive diseases that manifest later in life. As smokers develop these problems, smoking behavior and biomarkers of harm may be affected therefore we will restrict enrollment to those under age 65
14. provide baseline CO reading less than 10 at initial session
15. current use (or use within past 14 days) of any medication that affects the biotransformation of nicotine, such as anticonvulsant drugs, rifampin, and disulfiram; or any psychoactive medications which can affect smoking behaviors.
16. any conditions viewed by the PI or study physician as creating a potential increased risk to a participant due to their participation will be reasons for exclusion
17. at the discretion of the PI, any participants viewed as non-compliant will be excluded from further participation
18. Smoke cigarettes with a filter size other than standard or slim sized as the topography mouthpieces are sized for standard filters and have an adapter for slim cigarettes only.
19. Participants with a positive breath alcohol reading at intake session where they are being consented may be rescheduled. If participants have a positive breath alcohol at a rescheduled intake session, they will be excluded.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2012-12; Primary Completion 2014-10 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Number of cigars consumed daily | 20 days
  The number of cigars smoked each day.

SECONDARY OUTCOMES:
Carbon monoxide measurements | Each study day 0, 5, 10, 15, 20
Nicotine metabolites from urine samples | 20 days
  Measures of NNK, mercapturic acid metabolites, total nicotine equivalents.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Strasser, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be made publicly available via a request to study PI within one year of completion of the study.